CLINICAL TRIAL: NCT02180217
Title: Phase III, Multi-center, Double-blind, Randomized Withdrawal Study of LCI699 Following a 24 Week, Single-arm, Open-label Dose Titration and Treatment Period to Evaluate the Safety and Efficacy of LCI699 for the Treatment of Patients With Cushing's Disease
Brief Title: Safety and Efficacy of LCI699 for the Treatment of Patients With Cushing's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCI699C2301; 2013-004766-34 (EudraCT Number)
Record Dates: First submitted 2014-06-17; First posted 2014-07-02 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Cushings Disease
Keywords: LCI699; osilodrostat; Cushings Disease; open-label dose titration; randomized withdrawal
MeSH Terms: conditions — Adrenocortical Hyperfunction | interventions — Osilodrostat

STUDY DESIGN:
Intervention Model Description: It is a double-blind, randomized withdrawal study of LCI699 following a 24 week, single-arm, open-label dose titration and treatment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- osilodrostat (LCI699) (Experimental): Consisted of a single-arm, open-label, osilodrostat dose-titration in individual patients and then osilodrostat during a double-blind, placebo controlled RW Period.
  Interventions: Drug: osilodrostat
- LCI699 Placebo (Placebo Comparator): Consisted of a single-arm, open-label, osilodrostat dose-titration in individual patients and then placebo during a double-blind, placebo controlled RW Period.
  Interventions: Drug: LCI699 matching placebo

INTERVENTIONS:
Drug: osilodrostat — Osilodrostat comes in the form of film-coated tablets for oral administration, in the following strengths: 1 mg, 5 mg, 10 mg, and 20 mg. The maximum dose of osilodrostat was 30 mg bid.
  Other Names: LCI699
  Arms: osilodrostat (LCI699)
Drug: LCI699 matching placebo — Osilodrostat placebo comes in the form of film-coated tablets for oral administration, in the following strengths: 1 mg, 5 mg, 10 mg, and 20 mg. The maximum dose of osilodrostat placebo was 30 mg bid.
  Arms: LCI699 Placebo

SUMMARY:
The study aimed to confirm long-term efficacy and safety of LCI699 for the treatment of patients with Cushing's disease. It was a pivotal trial which supported the registration of LCI699 for the treatment of patients with Cushing's disease in the US and the EU.

This is a phase lll, multi-center, double-blind, randomized withdrawal study of LCI699 following a 24 week, single-arm, open-label dose titration and treatment period which evaluated the safety and efficacy of LCI699 for the treatment of patients with Cushing's disease.

DETAILED DESCRIPTION:
The primary objective compared the complete response rate at the end of the 8-week period of randomized withdrawal (Week 34) between patients randomized to continued osilodrostat therapy vs.

placebo. The key secondary objective assessed the complete response rate at the end of individual dose titration and treatment with osilodrostat in the initial single-arm, open label period (Week 24).

Eligible patients were randomized in a double-blinded fashion at Week 26 at a 1:1 ratio either to continue treatment with osilodrostat at the same dose or to matching placebo. Randomization was stratified by osilodrostat dose at Week 24 (≤ 5mg bid vs. >5mg bid); and history of pituitary irradiation (yes/no).

The study had four periods combined in the Core Period (Study Period 1 to 4) and an optional Extension Period. The optional Extension Period starting at Week 48.

Study Period 1 consisted of a single-arm, open-label, osilodrostat dose-titration in individual patients (Week 1 to Week 12). Dose adjustments were based on the mean of three 24-hour UFC (mUFC) values as measured by the central laboratory.

During study Period 2 (Week 13 to Week 24), osilodrostat efficacy and safety were assessed at the therapeutic dose determined during study Period 1. Patients whose mUFC became elevated during this period had their osilodrostat dose increased further, if it was tolerated, up to 30 mg bid. Such patients were followed for long-term safety and efficacy and were not considered responders for the key secondary endpoint, hence were not randomized in Study Period 3.

Study Period 3 was a double-blind, placebo-controlled randomized withdrawal (RW) Period (Week 26 to Week 34). In order to be eligible for randomization in study Period 3, patients had to have completed dose titration during study Period 1, and had to be classified as complete responders at Week 24 of study Period 2. Patients not eligible for randomization received open-label osilodrostat until the end of the Core Period (Week 48), unless there was a reason to discontinue from the study prematurely.

During study Period 3, mUFC was measured at scheduled visits every 2 weeks. However, patients were also allowed to have unscheduled visits at any time during the RW if they reported symptoms of hypercortisolism or hypocortisolism.

The dose of study drug remained unchanged for patients who maintained a normal mUFC and did not develop adverse events (AEs) related to study drug during RW. The Investigator could reduce or temporally withhold a dose of study drug for safety reasons at any time during the study, including the RW Period.

During this study period, a patient was discontinued from the RW Period and declared a nonresponder, if the mUFC increased to >1.5×ULN. After discontinuation from RW treatment, or at the end of the RW Period (Week 34), whichever came first, the patient resumed open-label osilodrostat at a dose selected by the Investigator.

Patients who discontinued from the study during the RW Period were no longer in the study, and consequently were not permitted to receive open-label osilodrostat and could not move to study Period 4.

Patients who discontinued from RW treatment due to lack of efficacy resumed open-label osilodrostat at the time of discontinuation, which could occur before Week 34. Patients who were not discontinued during RW resumed open-label osilodrostat at the end of RW (Week 34) and continued osilodrostat thereafter (study Period 4).

The Novartis study team, the patient, the Investigator, and all other site staff remained blinded to treatment assignment from the time of randomization to the time of database lock at the end of the Core Period. Novartis Drug Supply Management department members were unblinded in order to prepare the study drug supplies.

Study Period 4 was a single-arm, open-label therapy (end of Week 34 to Week 48). At the end of Week 34, all patients received open-label osilodrostat treatment. The Investigator had the discretion to select the dose during this period.

Patients continued open-label therapy until Week 48. At Week 48, patients had the option to enter an Extension Period, or discontinue osilodrostat at Week 48 to conclude with an end of Core Period visit 4 weeks off study drug (at Week 52).

Patients who continued to receive clinical benefit, as assessed by the study Investigator, and who wished to enter the Extension Period were re-consented at Week 48. Patients entered the Extension period without interruption of study drug or assessments. At the end of the study, patients who continued to benefit from treatment were offered to participate in a separate long-term safety follow-up study. The optional Extension Period ended after all patients completed Week 72 or discontinued early.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female patients aged 18 - 75 years.
3. Patients must have confirmed Cushing's disease that is persistent or recurrent.
4. Patients with a history of prior pituitary surgery must be at least 30 days post-surgery to be eligible for inclusion in this study.
5. Patients that received glucocorticoid replacement therapy post-operatively must have discontinued such therapy for at least one week, or 5 half-lives, whichever is longer, prior to screening.
6. Patients with de novo Cushing's disease can be included only if they are not considered candidates for surgery.
7. Patients with a history of pituitary irradiation can be included, provided that at least 2 years (stereotactic radiosurgery) or 3 years (conventional radiation) have elapsed from the time of last radiation treatment to the time of enrollment into this study.
8. Patients are permitted to washout current drug therapy to meet these entry criteria if they have a known diagnosis of Cushing's disease.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half lives at the time of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
2. History of hypersensitivity to LCI699 or to drugs of similar chemical classes.
3. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
4. Patients with risk factors for QTc prolongation or Torsade de Pointes.
5. Pregnant or nursing (lactating) women.
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after completion of dosing.
7. Patients with compression of the optic chiasm due to a macroadenoma or patients at high risk of compression of the optic chiasm (tumor within 2 mm of optic chiasm).
8. Patients who have a known inherited syndrome as the cause for hormone over secretion.
9. Patients with Cushing's syndrome due to ectopic ACTH secretion or ACTH-independent (adrenal) Cushing's syndrome.
10. Patients who have undergone major surgery within 1 month prior to screening.
11. Hypertensive patients with uncontrolled blood pressure.
12. Diabetic patients with poorly controlled diabetes.
13. Patients who are not euthyroid as judged by the investigator.
14. Patients who have a history of: congestive heart failure, unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, acute MI less than one year prior to study entry, or clinically significant impairment in cardiovascular function.
15. Patients with moderate to severe renal impairment.
16. Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with defined elevated ALT/ AST/ Bilirubin.
17. Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator or the sponsor's medical monitor.
18. Patients who have a history of alcohol or drug abuse in the 6 month period prior to study treatment.
19. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- United States (12):
  - University of Colorado Hospital SC - LCI699C2301, Aurora, Colorado
  - Emory University School of Medicine G2304 - C2301, Atlanta, Georgia
  - Northwestern University SC - LCI699C2301, Chicago, Illinois
  - The Johns Hopkins University School of Medicine Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital Neuroendocrine Unit, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mount Sinai School of Medicine SC - LCI699C2301, New York, New York
  - Columbia University Medical Center New York Presbyterian SC - LCI699C2301, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University SC LCI699C2301, Portland, Oregon
  - University of Pennsylvania Clinical Studies Unit Unniv SC, Philadelphia, Pennsylvania
  - Medical College of Wisconsin MCW 2, Milwaukee, Wisconsin
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (4):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (3):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Cali, Colombia
- France (5):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
- Germany (2):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, München
- India (4):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Chandigarh, Punjab
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, New Delhi
- Italy (7):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Napoli
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Songkhla, Thailand
- Novartis Investigative Site, Istanbul, TUR, Turkey (Türkiye)
- Novartis Investigative Site, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fleseriu M, Pivonello R, Lacroix A, Biller BMK, Feelders R, Gadelha M, Bertherat J, Belaya Z, Piacentini A, Pedroncelli AM, Newell-Price J. Osilodrostat dose impact on efficacy/safety in Cushing's disease: large, pooled analysis of LINC 2, 3, and 4. Eur J Endocrinol. 2025 Oct 30;193(5):606-617. doi: 10.1093/ejendo/lvaf207. PMID 41052284
- [Derived] Newell-Price J, Fleseriu M, Pivonello R, Feelders RA, Gadelha MR, Lacroix A, Witek P, Heaney AP, Piacentini A, Pedroncelli AM, Biller BMK. Improved Clinical Outcomes During Long-term Osilodrostat Treatment of Cushing Disease With Normalization of Late-night Salivary Cortisol and Urinary Free Cortisol. J Endocr Soc. 2024 Nov 12;9(1):bvae201. doi: 10.1210/jendso/bvae201. eCollection 2024 Nov 26. PMID 39610378
- [Derived] Pivonello R, Fleseriu M, Newell-Price J, Shimatsu A, Feelders RA, Kadioglu P, Tabarin A, Brue TC, Geer EB, Piacentini A, Pedroncelli AM, Biller BMK. Improvement in clinical features of hypercortisolism during osilodrostat treatment: findings from the Phase III LINC 3 trial in Cushing's disease. J Endocrinol Invest. 2024 Oct;47(10):2437-2448. doi: 10.1007/s40618-024-02359-6. Epub 2024 May 2. PMID 38696122
- [Derived] Gadelha M, Snyder PJ, Witek P, Bex M, Belaya Z, Turcu AF, Feelders RA, Heaney AP, Paul M, Pedroncelli AM, Auchus RJ. Long-term efficacy and safety of osilodrostat in patients with Cushing's disease: results from the LINC 4 study extension. Front Endocrinol (Lausanne). 2023 Aug 23;14:1236465. doi: 10.3389/fendo.2023.1236465. eCollection 2023. PMID 37680892
- [Derived] Fontaine-Sylvestre C, Letourneau-Guillon L, Moumdjian RA, Berthelet F, Lacroix A. Corticotroph tumor progression during long-term therapy with osilodrostat in a patient with persistent Cushing's disease. Pituitary. 2021 Apr;24(2):207-215. doi: 10.1007/s11102-020-01097-1. Epub 2020 Oct 19. PMID 33074401
- [Derived] Pivonello R, Fleseriu M, Newell-Price J, Bertagna X, Findling J, Shimatsu A, Gu F, Auchus R, Leelawattana R, Lee EJ, Kim JH, Lacroix A, Laplanche A, O'Connell P, Tauchmanova L, Pedroncelli AM, Biller BMK; LINC 3 investigators. Efficacy and safety of osilodrostat in patients with Cushing's disease (LINC 3): a multicentre phase III study with a double-blind, randomised withdrawal phase. Lancet Diabetes Endocrinol. 2020 Sep;8(9):748-761. doi: 10.1016/S2213-8587(20)30240-0. Epub 2020 Jul 27. PMID 32730798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 132 patients were planned, 137 were enrolled and 137 were analyzed.
Groups:
- Non-randomized: All participants in this group took open label osilodrostat, before and after randomization.
Period: Overall Study
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Started | 36 | 35 | 66
Discontinued at/Prior to Week 12 (W12) | 0 | 0 | 7
Discont. at/Prior to W26 But After W12 | 0 | 0 | 12
Discontinued Prior to W48 But After W26 | 0 | 2 | 3
Completed Week 48 (Core Phase) | 36 | 33 | 44
Completed W48, Did Not Enter Ext. Phase | 1 | 3 | 3
Completed W48, Entered Ext. Phase | 35 | 30 | 41
Discontinued Extension Phase | 12 | 6 | 16
Completed Ext. Phase | 23 | 24 | 25
Completed (Completed = Completed Core/Extension Phase) | 24 | 27 | 28
Not Completed | 12 | 8 | 38
Not completed — Adverse Event | 3 | 2 | 22
Not completed — Death | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Subject/Guardian decision | 5 | 3 | 6
Not completed — Physician Decision | 1 | 1 | 6
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized | Total
Number analyzed (Participants) | 36 | 35 | 66 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.27) | 42.0 (13.47) | 39.0 (13.38) | 41.2 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 54 | 106
  Male | 6 | 13 | 12 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 27 | 23 | 39 | 89
  Black | 0 | 3 | 1 | 4
  Asian | 7 | 7 | 25 | 39
  Other | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Primary Efficacy Responder at Week 34 by Randomized Treatment and Strata
Description: To compare the complete response rate at the end of the 8-week period of randomized withdrawal between randomized patients.A primary efficacy responder is defined as a randomized patient who has mUFC ≤ ULN at Week 34 and who was neither discontinued (study or RW treatment) nor had osilodrostat dose increase above the level at Week 26 during the RW Period of the study. mUFC: mean urinary free cortisol; ULN: Upper Limit of Normal
Time Frame: Week 34 (8 weeks)
Population: Randomized analysis set (RAS): comprises all randomized patients who received at least one dose of randomized drug (osilodrostat or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo
Number analyzed (Participants) | 36 | 34
Percentage of participants | 86.1 | 29.4
Statistical Analysis 1: Comparison: Osilodrostat (LCI699) vs LCI699 Placebo; Test type: Other; p < .001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 13.71, 95% CI 2-sided [3.73 to 53.44]

2. Secondary Outcome: Percentage of Secondary Efficacy Responder at Week 24 (Key Secondary Endpoint)
Description: To assess the complete response rate at the end of individual dose-titration and treatment with LCI699 in the initial single-arm, open label period. A Key secondary efficacy responder is defined as a patient in FAS who has mUFC ≤ ULN at Week 24 and the dose of osilodrostat during Study Period 2 (Weeks 13-24) was not increased above the level established at the end of Study Period 1 (Week 12). Patients who had missing mUFC assessment at Week 24 will be counted as non-responders for the key secondary endpoint.
Time Frame: Week 24
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: Consisted of all participants who were enrolled and treated in the open label osilodrostat.
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 52.6 [43.9 to 61.1]

3. Secondary Outcome: Time-to-loss of Control of Mean Urinary Free Cortisol (mUFC) by Randomized Treatment Group
Description: Time-to-loss of control of mUFC during the RW Period, defined as the time (in days) from randomization to the first evidence of loss of control (defined as mUFC assessment >1.5 ULN based on central laboratory result & at least 2 of the associated individual urine samples showing UFC >1.5×ULN) within the RW period. A patient without evidence of loss of control was censored at the date of the last assessment with mUFC ≤ 1.5 ULN. If a patient discontinued randomized treatment without having a UFC assessment, they were censored at the date of randomization. The measure type (number) refers to an Event probability estimate 8 weeks after randomization.
Time Frame: 8 weeks after randomization
Population: Randomized analysis set (RAS): comprised all randomized patients who received at least one dose of randomized drug (osilodrostat or placebo).
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo
Number analyzed (Participants) | 36 | 34
Percentage | 5.6 [1.4 to 20.4] | 61.1 [45.0 to 77.5]

4. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate is defined as percentage of enrolled participants with mUFC ≤ ULN
Time Frame: Week 12, Week 24, Week 48, Week 72, last observed value
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Percentage of participants
  Week 12 | 86.1 | 91.4 | 53.0
  Week 24 | 100.0 | 97.1 | 34.8
  Week 48 | 88.9 | 77.1 | 48.5
  Week 72: number analyzed (Participants) | 35 | 30 | 41
  Week 72 | 82.9 | 83.3 | 78.0
  Last observed value | 69.4 | 74.3 | 53.0

5. Secondary Outcome: Actual Change From Baseline in mUFC
Description: Actual change in mUFC from baseline.
Time Frame: Weeks 12, 24, 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: nmol/24h
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
nmol/24h
  Actual Baseline (BL) | 890.0 (1275.66) | 560.0 (548.84) | 1305.8 (2012.21)
  Wk 12: Act. change from BL: number analyzed (Participants) | 33 | 34 | 58
  Wk 12: Act. change from BL | -848.4 (1335.66) | -510.3 (556.84) | -1021.3 (1825.55)
  Wk 24: Act. change from BL: number analyzed (Participants) | 36 | 35 | 54
  Wk 24: Act. change from BL | -821.2 (1283.03) | -485.5 (558.99) | -930.3 (1778.04)
  Wk 48: Act. change from BL: number analyzed (Participants) | 34 | 32 | 42
  Wk 48: Act. change from BL | -708.2 (983.14) | -477.1 (529.04) | -1189.9 (2042.48)
  Wk 72: Act. change from BL: number analyzed (Participants) | 32 | 29 | 35
  Wk 72: Act. change from BL | -680.7 (1003.63) | -536.7 (585.78) | -826.7 (1684.92)
  Last avail. assess.: Act. change from BL | -795.2 (1286.22) | -387.3 (605.63) | -893.4 (1969.56)

6. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Fasting Glucose
Description: Actual change in fasting glucose from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
mg/dL
  Baseline: number analyzed (Participants) | 34 | 33 | 62
  Baseline | 102.7 (35.23) | 90.5 (18.53) | 101.8 (31.00)
  Wk 48: number analyzed (Participants) | 33 | 30 | 38
  Wk 48 | -7.9 (32.24) | -5.5 (12.13) | -14.1 (22.66)
  Wk 72: number analyzed (Participants) | 30 | 25 | 32
  Wk 72 | -0.5 (16.84) | -4.4 (15.13) | -10.8 (24.02)
  Last avail. assessment: number analyzed (Participants) | 34 | 32 | 62
  Last avail. assessment | -8.6 (37.05) | -0.6 (21.00) | -15.6 (26.62)

7. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Hemoglobin A1C (HbA1C)
Description: Actual change in glycosylated hemoglobin (HbA1c) from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
percentage
  Baseline | 6.1 (0.98) | 5.8 (0.93) | 6.0 (0.97)
  Wk 48: number analyzed (Participants) | 35 | 33 | 42
  Wk 48 | -0.3 (0.86) | -0.4 (0.56) | -0.4 (0.65)
  Wk 72: number analyzed (Participants) | 33 | 29 | 35
  Wk 72 | -0.4 (0.66) | -0.4 (0.47) | -0.4 (0.64)
  Last avail. assessment | -0.3 (0.78) | -0.2 (0.47) | -0.3 (0.68)

8. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Cholesterol, LDL Cholesterol, HDL Cholesterol & Triglyceride
Description: Actual change in Cholesterol, LDL Cholesterol, HDL Cholesterol & Triglyceride from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
mmol/L
  Cholesterol: BL: number analyzed (Participants) | 36 | 34 | 66
  Cholesterol: BL | 5.5 (1.22) | 5.3 (0.90) | 5.1 (1.24)
  Cholesterol: Wk 48: number analyzed (Participants) | 35 | 32 | 41
  Cholesterol: Wk 48 | -0.7 (0.87) | -0.4 (0.89) | -0.5 (0.90)
  Cholesterol: Wk 72: number analyzed (Participants) | 33 | 27 | 33
  Cholesterol: Wk 72 | -0.4 (0.96) | -0.3 (0.75) | -0.4 (0.98)
  Cholesterol: Last avail. assessment: number analyzed (Participants) | 36 | 34 | 66
  Cholesterol: Last avail. assessment | -0.3 (1.16) | -0.3 (1.03) | -0.4 (1.15)
  LDL Cholesterol: BL: number analyzed (Participants) | 36 | 34 | 66
  LDL Cholesterol: BL | 3.2 (1.09) | 3.1 (0.77) | 2.9 (0.94)
  LDL Cholesterol: Wk 48: number analyzed (Participants) | 35 | 32 | 40
  LDL Cholesterol: Wk 48 | -0.3 (0.75) | -0.2 (0.74) | -0.1 (0.82)
  LDL Cholesterol: Wk 72: number analyzed (Participants) | 33 | 27 | 33
  LDL Cholesterol: Wk 72 | -0.2 (0.77) | -0.2 (0.66) | -0.1 (0.86)
  LDL Cholesterol: Last avail asses: number analyzed (Participants) | 36 | 34 | 65
  LDL Cholesterol: Last avail asses | -0.1 (0.98) | -0.2 (0.88) | -0.1 (0.99)
  HDL Cholesterol: BL: number analyzed (Participants) | 36 | 34 | 66
  HDL Cholesterol: BL | 1.7 (0.55) | 1.5 (0.36) | 1.6 (0.42)
  HDL Cholesterol: Wk 48: number analyzed (Participants) | 35 | 32 | 41
  HDL Cholesterol: Wk 48 | -0.3 (0.39) | -0.2 (0.17) | -0.3 (0.28)
  HDL Cholesterol: Wk 72: number analyzed (Participants) | 33 | 27 | 33
  HDL Cholesterol: Wk 72 | -0.2 (0.39) | -0.2 (0.27) | -0.3 (0.28)
  HDL Cholesterol: Last avail assess: number analyzed (Participants) | 36 | 34 | 66
  HDL Cholesterol: Last avail assess | -0.2 (0.40) | -0.1 (0.27) | -0.2 (0.34)
  Triglyceride: BL: number analyzed (Participants) | 36 | 34 | 66
  Triglyceride: BL | 1.5 (0.78) | 1.4 (0.62) | 1.6 (1.74)
  Triglyceride: Wk 48: number analyzed (Participants) | 35 | 32 | 41
  Triglyceride: Wk 48 | -0.1 (0.49) | 0.0 (0.54) | 0.0 (1.22)
  Triglyceride: Wk 72: number analyzed (Participants) | 33 | 28 | 33
  Triglyceride: Wk 72 | 0.0 (0.57) | -0.1 (0.67) | 0.0 (0.60)
  Triglyceride: Last avail. assess: number analyzed (Participants) | 36 | 34 | 66
  Triglyceride: Last avail. assess | 0.0 (0.64) | -0.1 (0.75) | 0.1 (1.48)

9. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Sitting Systolic Blood Pressure (SBP) & Sitting Diastolic Blood Pressure (DBP)
Description: Actual change in sitting SBP & DBP from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
mmHg
  SBP: Baseline | 132.2 (15.44) | 128.8 (11.93) | 134.0 (16.34)
  SBP: Wk 48: number analyzed (Participants) | 35 | 33 | 43
  SBP: Wk 48 | -15.2 (17.00) | -4.8 (12.28) | -9.2 (15.48)
  SBP: Wk 72: number analyzed (Participants) | 34 | 29 | 36
  SBP: Wk 72 | -12.2 (15.90) | -8.2 (19.41) | -9.4 (19.08)
  SBP: Last avail. assessment | -8.2 (15.25) | -4.6 (15.20) | -10.8 (15.31)
  DBP: Baseline | 85.3 (11.38) | 85.0 (10.03) | 85.4 (10.53)
  DBP: Wk 48: number analyzed (Participants) | 35 | 33 | 43
  DBP: Wk 48 | -7.8 (11.63) | -5.1 (9.66) | -6.0 (11.79)
  DBP: Wk 72: number analyzed (Participants) | 34 | 29 | 36
  DBP: Wk 72 | -5.9 (11.17) | -7.0 (10.33) | -4.8 (12.26)
  DBP: Last avail. assessment | -3.4 (11.79) | -3.5 (11.50) | -5.0 (10.45)

10. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Weight
Description: Actual change in weight from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
kg
  Baseline | 78.2 (19.02) | 83.4 (24.73) | 80.7 (23.06)
  Wk 48: number analyzed (Participants) | 36 | 33 | 43
  Wk 48 | -3.4 (5.64) | -3.9 (5.77) | -4.0 (5.82)
  Wk 72: number analyzed (Participants) | 34 | 29 | 36
  Wk 72 | -3.7 (6.93) | -5.0 (6.03) | -5.6 (6.75)
  Last avail. assessment | -2.9 (8.28) | -3.7 (11.13) | -4.2 (6.35)

11. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Body Mass Index (BMI)
Description: Actual change in BMI from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
kg/m^2
  Baseline | 29.6 (7.36) | 30.9 (8.38) | 30.4 (7.74)
  Wk 48: number analyzed (Participants) | 36 | 33 | 43
  Wk 48 | -1.3 (2.22) | -1.5 (2.12) | -1.5 (2.17)
  Wk 72: number analyzed (Participants) | 34 | 29 | 36
  Wk 72 | -1.4 (2.79) | -1.8 (2.14) | -2.0 (2.55)
  Last avail. assessment | -1.2 (3.34) | -1.5 (3.94) | -1.6 (2.41)

12. Secondary Outcome: Actual Change From Baseline in Cardiovascular-related Parameter Associated With Cushing's Disease: Waist Circumference
Description: Actual change in waist circumference from baseline.
Time Frame: Baseline, Weeks 48, 72, last available assessment
Population: Full analysis set (FAS): comprises all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
cm
  Baseline: number analyzed (Participants) | 35 | 33 | 65
  Baseline | 100.5 (16.81) | 103.7 (18.26) | 105.0 (21.15)
  Wk 48: number analyzed (Participants) | 34 | 32 | 43
  Wk 48 | -5.1 (6.26) | -4.2 (10.12) | -4.7 (7.07)
  Wk 72: number analyzed (Participants) | 33 | 29 | 36
  Wk 72 | -5.1 (7.18) | -6.1 (9.86) | -7.4 (8.53)
  Last avail. assessment: number analyzed (Participants) | 35 | 33 | 65
  Last avail. assessment | -4.7 (10.05) | -5.2 (12.24) | -6.2 (9.96)

13. Secondary Outcome: Actual Change From Baseline in Patient-Reported Outcomes (Cushing's Health-Related Quality of Life (QoL)) - Total Score
Description: Cushing's Disease Health-Related Quality of Life Questionnaire was developed to evaluate quality of life in patients with Cushing's syndrome. It is comprised of 12 items that capture patient responses on 7 concepts: daily activities, healing & pain, mood & self-confidence, social concerns, physical appearance, memory & concern about the future. These items are measured on a 5- point Likert-type scale assessing how often or how much each item has been related to the patient's Cushing's disease in the previous 4 weeks. The raw score is calculated by summing the individual item scores prior to being standardized so that the total score ranges from 0 to 100. Content reliability, sensitivity to change & psychometric properties have been validated in patients with Cushing's disease. Patients were asked to complete the questionnaire prior to clinical assessments being undertaken. Increases from baseline are indicative of an improvement.
Time Frame: Baseline, Week (W) 48, W72, Last available assessment
Population: FAS: Comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
scores on a scale
  Baseline | 44.4 (18.33) | 43.2 (22.45) | 40.5 (17.61)
  Week 48: number analyzed (Participants) | 35 | 32 | 43
  Week 48 | 16.1 (15.15) | 10.2 (16.57) | 13.2 (17.79)
  Week 72: number analyzed (Participants) | 32 | 28 | 37
  Week 72 | 15.8 (16.08) | 12.6 (20.68) | 16.3 (21.31)
  Last available assess.: number analyzed (Participants) | 36 | 35 | 65
  Last available assess. | 16.1 (15.99) | 11.8 (20.51) | 12.9 (18.91)

14. Secondary Outcome: Actual Change From Baseline in Patient-Reported Outcomes: Beck Depression Inventory-II (BDI-II)
Description: BDI-II is a patient-reported instrument developed to measure the severity of depression in adults & adolescents aged 13 years & older. It is designed to be completed by the patient on paper & takes approximately 5 minutes to complete. The BDI-II consists of 21 items designed to assess the intensity of depression in clinical & normal patients in the preceding 2 weeks. Items are rated on a 4-point severity scale of 0 ('not at all') to 3 ('extreme' form of each symptom) with differing response options for each item. A global score ranging from 0 to 63 is calculated with a higher score representing a greater level of depression. The following scoring guidelines for interpretation of BDI-II have been suggested (Smarr, 2011): Minimal range =0-13, Mild depression =14-19, Moderate depression =20-28 and Severe depression = 29-63. Patients were asked to complete the questionnaire prior to clinical assessments being undertaken. A reduction from baseline in BDI-II is indicative of an improvement.
Time Frame: Baseline, W48, W72, Last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: scores on a a scale
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
scores on a a scale
  Baseline | 15.1 (11.14) | 17.8 (9.93) | 17.3 (10.67)
  W48: number analyzed (Participants) | 35 | 32 | 43
  W48 | -4.8 (9.84) | -5.3 (7.99) | -7.0 (10.17)
  W72: number analyzed (Participants) | 32 | 28 | 36
  W72 | -6.0 (9.55) | -4.6 (9.41) | -9.0 (12.34)
  Last avail. assess.: number analyzed (Participants) | 36 | 35 | 65
  Last avail. assess. | -6.2 (9.93) | -5.0 (9.49) | -4.9 (10.66)

15. Secondary Outcome: Actual Change in Patient-Reported Outcomes: EQ-5D-5L Utility Index
Description: The EQ-5D-5L questionnaire is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. It is cognitively undemanding, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire. The EQ-5D-5L measures 5 items on mobility, self-care, usual activities, pain/discomfort, anxiety/depression, measured on 5 levels: no problems, slight problems, moderate problems, severe problems, & extreme problems. A utility index can be computed from the EQ 5D-5L descriptive system with utility scores ranging from -0.281 (worst imaginable health state) to 1 (best imaginable health state), with -0.281 representing an "unconscious" health state. A single index value is analyzed for the EQ-5D-5L score. An increase from baseline in the EQ-ED-5L utility index is indicative of an improvement.
Time Frame: Baseline, W48, W72, Last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Scores on a scale
  Baseline | 0.7 (0.24) | 0.7 (0.24) | 0.7 (0.28)
  Week 48: number analyzed (Participants) | 35 | 32 | 43
  Week 48 | 0.1 (0.18) | 0 (0.25) | 0.1 (0.18)
  Week 72: number analyzed (Participants) | 32 | 28 | 36
  Week 72 | 0.1 (0.18) | 0.1 (0.26) | 0.1 (0.19)
  Last avail. assess.: number analyzed (Participants) | 36 | 35 | 65
  Last avail. assess. | 0.1 (0.22) | 0 (0.28) | 0.1 (0.23)

16. Secondary Outcome: Actual Change in Patient-Reported Outcomes: EQ-5D-5L Vascular Analog Scale (VAS)
Description: The EQ-5D-5L also includes a 20 cm vertical, VAS (visual analogue scale) with on a scale of 0-100, with endpoints labeled 100 = 'the best health you can imagine' and 0 = 'the worst health you can imagine'. A single index value is analyzed for the VAS score. An increase from baseline in the EQ-ED-5L VAS is indicative of an improvement.
Time Frame: Baseline, W48, W72, Last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Scores on a scale
  Baseline | 61.3 (18.97) | 64.2 (16.37) | 60.8 (21.09)
  Week 48: number analyzed (Participants) | 35 | 31 | 43
  Week 48 | 12.6 (20.64) | 6.9 (12.56) | 9.7 (17.16)
  Week 72: number analyzed (Participants) | 32 | 27 | 36
  Week 72 | 11.2 (18.98) | 6.6 (15.47) | 10.1 (19.80)
  Last avail. assess.: number analyzed (Participants) | 36 | 34 | 65
  Last avail. assess. | 12.1 (19.71) | 6.4 (18.65) | 6.2 (20.42)

17. Secondary Outcome: Change From Baseline in the Physical Features of Cushing's Disease by Photography
Description: Improvement from baseline to Weeks 48, 72 and End of Treatment (Extension period) in each of the following clinical signs of Cushing's disease by photography: facial rubor, hirsutism, striae, supraclavicular fat pad, dorsal fat pad, proximal muscle wasting (atrophy), central (abdominal) obesity, and ecchymoses (bruises).
Time Frame: Week 48, Week 72, Last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Percentage of participants
  W48: Facial rubor: number analyzed (Participants) | 30 | 30 | 37
  W48: Facial rubor | 50.0 [31.3 to 68.7] | 46.7 [28.3 to 65.7] | 43.2 [27.1 to 60.5]
  W48: Striae: number analyzed (Participants) | 30 | 30 | 37
  W48: Striae | 30.0 [14.7 to 49.4] | 23.3 [9.9 to 42.3] | 40.5 [24.8 to 57.9]
  W48:Supraclavicular fat pad: number analyzed (Participants) | 30 | 30 | 37
  W48:Supraclavicular fat pad | 56.7 [37.4 to 74.5] | 43.3 [25.5 to 62.6] | 54.1 [36.9 to 70.5]
  W48: Dorsal fat pad: number analyzed (Participants) | 30 | 30 | 37
  W48: Dorsal fat pad | 60.0 [40.6 to 77.3] | 40.0 [22.7 to 59.4] | 56.8 [39.5 to 72.9]
  W48: Proximal muscle atrophy: number analyzed (Participants) | 30 | 30 | 37
  W48: Proximal muscle atrophy | 40.0 [22.7 to 59.4] | 26.7 [12.3 to 45.9] | 45.9 [29.5 to 63.1]
  W48: Central obesity: number analyzed (Participants) | 30 | 30 | 37
  W48: Central obesity | 43.3 [25.5 to 62.6] | 30.0 [14.7 to 49.4] | 51.4 [34.4 to 68.1]
  W48: Ecchymoses: number analyzed (Participants) | 30 | 30 | 37
  W48: Ecchymoses | 33.3 [17.3 to 52.8] | 26.7 [12.3 to 45.9] | 43.2 [27.1 to 60.5]
  W72: Facial rubor: number analyzed (Participants) | 29 | 27 | 30
  W72: Facial rubor | 48.3 [29.4 to 67.5] | 55.6 [35.3 to 74.5] | 53.3 [34.3 to 71.7]
  W72: Striae: number analyzed (Participants) | 29 | 27 | 30
  W72: Striae | 27.6 [12.7 to 47.2] | 25.9 [11.1 to 46.3] | 36.7 [19.9 to 56.1]
  W72:Supraclavicular fat pad: number analyzed (Participants) | 29 | 27 | 30
  W72:Supraclavicular fat pad | 55.2 [35.7 to 73.6] | 51.9 [31.9 to 71.3] | 53.3 [34.3 to 71.1]
  W72: Dorsal fat pad: number analyzed (Participants) | 29 | 27 | 30
  W72: Dorsal fat pad | 69.0 [49.2 to 84.7] | 48.1 [28.7 to 68.1] | 53.3 [34.3 to 71.7]
  W72: Proximal muscle atrophy: number analyzed (Participants) | 29 | 27 | 30
  W72: Proximal muscle atrophy | 31.0 [15.3 to 50.8] | 25.9 [11.1 to 46.3] | 46.7 [28.3 to 65.7]
  W72: Central obesity: number analyzed (Participants) | 29 | 27 | 30
  W72: Central obesity | 37.9 [20.7 to 57.7] | 37.0 [19.4 to 57.6] | 43.3 [25.5 to 62.6]
  W72: Ecchymoses: number analyzed (Participants) | 29 | 27 | 30
  W72: Ecchymoses | 27.6 [12.7 to 47.2] | 29.6 [13.8 to 50.2] | 36.7 [19.9 to 56.1]
  End of Trial (EOT):Facial rubor: number analyzed (Participants) | 25 | 23 | 26
  End of Trial (EOT):Facial rubor | 60.0 [38.7 to 78.9] | 56.5 [34.5 to 76.8] | 53.8 [33.4 to 73.4]
  EOT: Striae: number analyzed (Participants) | 25 | 23 | 26
  EOT: Striae | 32.0 [14.9 to 53.5] | 34.8 [16.4 to 57.3] | 30.8 [14.3 to 51.8]
  EOT:Supraclavicular fat pad: number analyzed (Participants) | 25 | 23 | 26
  EOT:Supraclavicular fat pad | 52.0 [31.3 to 72.2] | 43.5 [23.2 to 65.5] | 42.3 [23.4 to 63.1]
  EOT: Dorsal fat pad: number analyzed (Participants) | 25 | 23 | 26
  EOT: Dorsal fat pad | 56.0 [34.9 to 75.6] | 52.2 [30.6 to 73.2] | 46.2 [26.6 to 66.6]
  EOT: Proximal muscle atrophy: number analyzed (Participants) | 25 | 23 | 26
  EOT: Proximal muscle atrophy | 36.0 [18.0 to 57.5] | 21.7 [7.5 to 43.7] | 50.0 [29.9 to 70.1]
  EOT: Central obesity: number analyzed (Participants) | 25 | 23 | 26
  EOT: Central obesity | 40.0 [21.1 to 61.3] | 39.1 [19.7 to 61.5] | 38.5 [20.0 to 59.4]
  EOT: Ecchymoses: number analyzed (Participants) | 25 | 23 | 26
  EOT: Ecchymoses | 28.0 [12.1 to 49.4] | 39.1 [19.7 to 61.5] | 38.5 [20.2 to 59.4]

18. Secondary Outcome: Change From Baseline in Bone Mineral Density - All Participants
Description: Actual change from baseline to Week 48 and the LOV in bone mineral density as measured by DXA scan at the lumbar spine and total hip. An increase in bone mineral density is indicative of an improvement..
Time Frame: Baseline, Week 48, Last observed value (LOV)
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Mean (Standard Error); unit: g/cm2
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
g/cm2
  Baseline (L1-L4 Lumbar Spine): number analyzed (Participants) | 28 | 27 | 58
  Baseline (L1-L4 Lumbar Spine) | 1.0 (0.20) | 1.0 (0.17) | 1.0 (0.18)
  W48 (L1-L4 Lumbar Spine): number analyzed (Participants) | 23 | 23 | 35
  W48 (L1-L4 Lumbar Spine) | 1.0 (0.19) | 1.0 (0.17) | 1.0 (0.19)
  LOV (L1-L4 Lumbar Spine): number analyzed (Participants) | 26 | 24 | 46
  LOV (L1-L4 Lumbar Spine) | 1.0 (0.20) | 1.0 (0.18) | 1.0 (0.18)
  Baseline (Total Hip): number analyzed (Participants) | 29 | 26 | 58
  Baseline (Total Hip) | 0.9 (0.18) | 0.8 (0.15) | 0.9 (0.16)
  W48 (Total Hip): number analyzed (Participants) | 24 | 21 | 35
  W48 (Total Hip) | 0.9 (0.17) | 0.8 (0.14) | 0.9 (0.16)
  LOV (Total Hip): number analyzed (Participants) | 27 | 22 | 46
  LOV (Total Hip) | 0.9 (0.17) | 0.8 (0.13) | 0.9 (0.16)

19. Secondary Outcome: Time-to-escape
Description: Escape was defined as the time (in days) from the first mUFC ≤ ULN to the first mUFC results > 1.5 x ULN with at least 2 individual UFC results > 1.5 x ULN the loss happened beyond 12-week dose titration period. Participants randomized to placebo were not included in the analysis.
Time Frame: From the first mUFC ≤ ULN to the first mUFC results > 1.5 x ULN with at least 2 individual UFC results > 1.5 x ULN
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat. This is a subset of the FAS participants who met all the criteria for Escape. The placebo patients + patients that did not reach mUFC <= ULN at some stage during the study are excluded from the denominator.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- All Participants: Consisted of all participants in the study under osilodrostat treatment
Arm/Group | All Participants
Number analyzed (Participants) | 97
days | 546.0 [212.0 to 968.0]

20. Secondary Outcome: LCI699 Exposures
Description: To evaluate exposures of LCI699 in patients with Cushing's disease. Plasma concentrations (predose, 0.75 h, 1.5 h, and 4 h post-dose) of LCI699. These are the maximum number of PAS subjects analyzed for each incident dose.
Time Frame: from week 2 to 10 at Predose, 0.75h, 1.5h, and 4h post-dose
Population: Pharmacokinetics analysis set (PAS) consists of all enrolled patients who receive at least one dose of osilodrostat and have at least one evaluable post-dosing PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Osilodrostat (LCI699) 2 mg: Participants received 2mg of osilodrostat
- Osilodrostat (LCI699) 3 mg: Participants received 3mg of osilodrostat
- Osilodrostat (LCI699) 5 mg: Participants received 5 mg of osilodrostat
- Osilodrostat (LCI699) 7 mg: Participants received 7 mg of osilodrostat
Arm/Group | Osilodrostat (LCI699) 2 mg | Osilodrostat (LCI699) 3 mg | Osilodrostat (LCI699) 5 mg | Osilodrostat (LCI699) 7 mg
Number analyzed (Participants) | 132 | 39 | 105 | 24
ng/ml
  Week (Wk) 2: Predose: number analyzed (Participants) | 79 | 0 | 0 | 0
  Week (Wk) 2: Predose | 1.904 (110.4) |  |  |
  Wk 2: 0.75h: number analyzed (Participants) | 14 | 0 | 0 | 0
  Wk 2: 0.75h | 1.907 (132.5) |  |  |
  Wk 2: 1.5h: number analyzed (Participants) | 3 | 0 | 0 | 0
  Wk 2: 1.5h | 5.1 (62.7) |  |  |
  Wk 2: 4h: number analyzed (Participants) | 18 | 0 | 0 | 0
  Wk 2: 4h | 5.818 (66.3) |  |  |
  Wk 4: Predose: number analyzed (Participants) | 50 | 2 | 31 | 0
  Wk 4: Predose | 2.104 (108.0) | 2.898 (109.1) | 3.584 (126.3) |
  Wk 4: 0.75h: number analyzed (Participants) | 2 | 0 | 9 | 0
  Wk 4: 0.75h | 0.859 (254.3) |  | 7.091 (137.8) |
  Wk 4: 1.5h: number analyzed (Participants) | 2 | 0 | 1 | 0
  Wk 4: 1.5h | 8.737 (3.6) |  | 24.2 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |
  Wk 4: 4h: number analyzed (Participants) | 1 | 0 | 9 | 0
  Wk 4: 4h | 8.930 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |  | 15.985 (48.3) |
  Wk 6: Predose: number analyzed (Participants) | 17 | 3 | 46 | 2
  Wk 6: Predose | 2.037 (63.5) | 2.392 (285.6) | 5.087 (122.9) | 8.065 (8.6)
  Wk 6: 0.75h: number analyzed (Participants) | 1 | 0 | 5 | 0
  Wk 6: 0.75h | 3.110 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |  | 5.223 (229.4) |
  Wk 6: 1.5h: number analyzed (Participants) | 0 | 1 | 1 | 0
  Wk 6: 1.5h |  | 22.4 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 21.4 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |
  Wk 6: 4h: number analyzed (Participants) | 1 | 1 | 5 | 0
  Wk 6: 4h | 8.380 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 18.6 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 18.373 (36.5) |
  Wk 8: Predose: number analyzed (Participants) | 13 | 5 | 35 | 3
  Wk 8: Predose | 2.198 (108.9) | 4.061 (67.4) | 4.487 (106.9) | 6.718 (34.2)
  Wk 8: 0.75h: number analyzed (Participants) | 0 | 0 | 0 | 0
  Wk 8: 1.5h: number analyzed (Participants) | 1 | 1 | 0 | 1
  Wk 8: 1.5h | 10.8 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 20.4 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |  | 32.1 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient.
  Wk 8: 4h: number analyzed (Participants) | 1 | 0 | 0 | 1
  Wk 8: 4h | 6.65 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |  |  | 32 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient.
  Wk 10: Predose: number analyzed (Participants) | 10 | 9 | 29 | 6
  Wk 10: Predose | 1.862 (128.9) | 3.007 (64.8) | 4.704 (106.8) | 5.451 (93.1)
  Wk 10: 0.75h: number analyzed (Participants) | 0 | 1 | 0 | 1
  Wk 10: 0.75h |  | 6.7 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient. |  | 17.1 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient.
  Wk 10: 1.5h: number analyzed (Participants) | 1 | 1 | 1 | 0
  Wk 10: 1.5h | 12.1 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 18.3 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 34.2 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient |
  Wk 10: 4h: number analyzed (Participants) | 0 | 1 | 1 | 1
  Wk 10: 4h |  | 15.8 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 27.2 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient | 35.5 (NA) — NA: CV% geo-mean could not be calculated with just 1 patient

21. Secondary Outcome: Percentage of Participants With Complete Response Rate (CRR)
Description: Complete response rate is defined as percentage of enrolled participants with mUFC ≤ ULN.
Time Frame: Week 12, Week 24, Week 48, Week 72, last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Percentage of participants
  Week 12 | 6.1 | 91.4 | 53.0
  Week 24 | 100 | 97.1 | 34.8
  Week 48 | 88.9 | 77.1 | 48.5
  Week 72: number analyzed (Participants) | 35 | 30 | 41
  Week 72 | 82.9 | 83.3 | 78.0
  Last available assess. | 69.4 | 74.3 | 53.0

22. Secondary Outcome: Percentage of Participants With Partial Response Rate (PRR)
Description: Partial response rate is defined as percentage of enrolled participants with ≥ 50% reduction from baseline in mUFC, but mUFC>ULN)
Time Frame: Week 12, Week 24, Week 48, Week 72, last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Percentage of participants
  Week 12 | 2.8 | 5.7 | 24.2
  Week 24 | 0.0 | 0.0 | 30.3
  Week 48 | 5.6 | 11.4 | 10.6
  Week 72: number analyzed (Participants) | 35 | 30 | 41
  Week 72 | 8.6 | 13.3 | 2.4
  Last available assess. | 22.2 | 11.4 | 22.7

23. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: Overall response rate is defined as percentage of enrolled participants with mUFC ≤ ULN or at least 50% reduction from baseline.
Time Frame: Week 12, Week 24, Week 48, Week 72, last available assessment
Population: FAS comprised all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Osilodrostat (LCI699) | LCI699 Placebo | Non-randomized
Number analyzed (Participants) | 36 | 35 | 66
Percentage of participants
  Week 12 | 88.9 | 97.1 | 77.3
  Week 24 | 100 | 97.1 | 65.2
  Week 48 | 94.4 | 88.6 | 59.1
  Week 72: number analyzed (Participants) | 35 | 30 | 41
  Week 72 | 91.4 | 96.7 | 80.5
  Last available assess. | 91.7 | 85.7 | 75.8

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from first dose of study treatment until 30 days after the last dose administration, up to maximum duration of about 245.1 weeks.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus up to 30 days after the last dose administration.
Groups:
- Osilodrostat: Consisted of a single-arm, open-label, osilodrostat dose-titration in individual patients and then osilodrostat during a double-blind, placebo controlled RW Period.
- All Participants: Consisted of all participants who were enrolled and treated with open label osilodrostat.
Arm/Group | Osilodrostat | LCI699 Placebo | Non-randomized | All Participants
All-Cause Mortality (participants affected / at risk) | 1/36 | 1/35 | 0/66 | 2/137
Serious Adverse Events (participants affected / at risk) | 13/36 | 10/35 | 32/66 | 55/137
Other Adverse Events (participants affected / at risk) | 34/36 | 35/35 | 65/66 | 134/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=36) | LCI699 Placebo (N=35) | Non-randomized (N=66) | All Participants (N=137)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 6 | 8
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 3 | 4
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 2 | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 1
Pituitary infarction (Endocrine disorders) | 0 | 0 | 1 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 2
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 3 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 2 | 3
Keratitis fungal (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Malignant pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 4 | 6
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 3
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 3
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 3 | 3
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cystitis glandularis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=36) | LCI699 Placebo (N=35) | Non-randomized (N=66) | All Participants (N=137)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 6 | 15
Bundle branch block right (Cardiac disorders) | 0 | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 3 | 3 | 8
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 1 | 3
Adrenal insufficiency (Endocrine disorders) | 7 | 10 | 17 | 34
Glucocorticoid deficiency (Endocrine disorders) | 10 | 9 | 8 | 27
Dry eye (Eye disorders) | 2 | 0 | 2 | 4
Eye pruritus (Eye disorders) | 0 | 2 | 0 | 2
Photophobia (Eye disorders) | 0 | 2 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 8 | 15
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 3 | 9
Constipation (Gastrointestinal disorders) | 4 | 1 | 5 | 10
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 14 | 27
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 8 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 17 | 11 | 34 | 62
Toothache (Gastrointestinal disorders) | 2 | 0 | 3 | 5
Vomiting (Gastrointestinal disorders) | 7 | 5 | 21 | 33
Application site rash (General disorders) | 0 | 2 | 0 | 2
Asthenia (General disorders) | 11 | 5 | 11 | 27
Chest discomfort (General disorders) | 1 | 0 | 4 | 5
Chills (General disorders) | 1 | 3 | 2 | 6
Fatigue (General disorders) | 8 | 13 | 24 | 45
Gait disturbance (General disorders) | 2 | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 2 | 1 | 3
Malaise (General disorders) | 1 | 2 | 7 | 10
Oedema (General disorders) | 1 | 3 | 5 | 9
Oedema peripheral (General disorders) | 8 | 5 | 9 | 22
Pain (General disorders) | 2 | 3 | 1 | 6
Pyrexia (General disorders) | 4 | 3 | 13 | 20
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1 | 6 | 8
Cystitis (Infections and infestations) | 3 | 2 | 1 | 6
Folliculitis (Infections and infestations) | 1 | 2 | 0 | 3
Fungal skin infection (Infections and infestations) | 1 | 2 | 0 | 3
Gastroenteritis (Infections and infestations) | 4 | 3 | 5 | 12
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 3 | 2 | 5
Influenza (Infections and infestations) | 5 | 8 | 10 | 23
Nasopharyngitis (Infections and infestations) | 9 | 11 | 13 | 33
Sinusitis (Infections and infestations) | 3 | 1 | 4 | 8
Tooth abscess (Infections and infestations) | 2 | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 7 | 14
Urinary tract infection (Infections and infestations) | 6 | 4 | 14 | 24
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 4 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 5
11-deoxycortisol increased (Investigations) | 3 | 1 | 2 | 6
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 1 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 4
Blood cholesterol increased (Investigations) | 2 | 0 | 1 | 3
Blood corticotrophin increased (Investigations) | 8 | 6 | 14 | 28
Blood testosterone increased (Investigations) | 2 | 1 | 13 | 16
Cortisol decreased (Investigations) | 3 | 0 | 1 | 4
Cortisol free urine decreased (Investigations) | 8 | 2 | 1 | 11
Cortisol free urine increased (Investigations) | 6 | 1 | 1 | 8
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 2
Hormone level abnormal (Investigations) | 5 | 1 | 12 | 18
Lipase increased (Investigations) | 1 | 2 | 1 | 4
Low density lipoprotein increased (Investigations) | 2 | 0 | 1 | 3
Renin increased (Investigations) | 3 | 0 | 3 | 6
Weight decreased (Investigations) | 2 | 2 | 5 | 9
Weight increased (Investigations) | 1 | 2 | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 3 | 7 | 11 | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 11 | 17
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 1 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10 | 12 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 13 | 7 | 29
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 11 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 6 | 13
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 6 | 9
Amnesia (Nervous system disorders) | 2 | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 5 | 4 | 17 | 26
Headache (Nervous system disorders) | 11 | 7 | 32 | 50
Hypoaesthesia (Nervous system disorders) | 1 | 4 | 4 | 9
Memory impairment (Nervous system disorders) | 2 | 1 | 2 | 5
Migraine (Nervous system disorders) | 0 | 1 | 4 | 5
Paraesthesia (Nervous system disorders) | 1 | 4 | 0 | 5
Somnolence (Nervous system disorders) | 2 | 0 | 3 | 5
Anxiety (Psychiatric disorders) | 3 | 2 | 7 | 12
Depression (Psychiatric disorders) | 3 | 3 | 7 | 13
Insomnia (Psychiatric disorders) | 4 | 2 | 7 | 13
Irritability (Psychiatric disorders) | 1 | 1 | 4 | 6
Panic attack (Psychiatric disorders) | 0 | 2 | 0 | 2
Sleep disorder (Psychiatric disorders) | 2 | 0 | 5 | 7
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0 | 3
Menstruation irregular (Reproductive system and breast disorders) | 0 | 2 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 10 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7 | 14
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 7
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 9 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 7 | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 7 | 10
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5
Hirsutism (Skin and subcutaneous tissue disorders) | 4 | 3 | 5 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 9
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 7 | 13
Rash (Skin and subcutaneous tissue disorders) | 8 | 3 | 10 | 21
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 4
Hypertension (Vascular disorders) | 5 | 5 | 14 | 24
Hypotension (Vascular disorders) | 7 | 3 | 3 | 13
Varicose vein (Vascular disorders) | 2 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The first 12 weeks of the study consisted of an individual dose-titration period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT02180217/SAP_002.pdf
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02180217/Prot_003.pdf